CLINICAL TRIAL: NCT00121511
Title: The Effect of Efudex (5-fluorouracil) Treatment on Photoaged Skin
Brief Title: The Effect of Efudex Treatment on Photoaged Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Dana L. Sachs, MD, Professor of Dermatology, Medical School, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Derm 549; 2005-0368
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Photo-aging; Keratosis
Keywords: photoaging; Actinic Keratoses; Efudex; 5 fluorouracil
MeSH Terms: conditions — Keratosis; Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Efudex (5-fluorouracil)

SUMMARY:
The researchers propose that skin improvements may be seen following a course of Efudex, (5-fluorouracil), a FDA-approved topical therapy (applied directly to the skin). These improvements could be the result of both a reduction of actinic keratoses (small red horny growths or flesh-colored wartlike growths caused by overexposure to ultraviolet radiation or the sun) and improvement of sun-damaged skin.

In addition, this research study is being done to determine if the expression of p53, a tumor suppressor gene (its activity stops the formation of tumors), is decreased following Efudex treatment. Mutations (abnormal changes) in the gene, called p53, are associated with a certain type of skin cancer. In addition, p53-mutated genes are known to exist in non-cancerous sun-damaged skin. Thus, the presence of p53 mutations may serve as a marker for both sun damage and an elevated risk of developing skin cancer.

DETAILED DESCRIPTION:
Efudex (5-fluorouracil) has been used as topical chemotherapy for the treatment of actinic keratoses (AKs) since the 1950's. Through many years of use, Efudex has been deemed to be a safe and effective therapy. It requires, however, a high level of patient compliance and is known to cause a vigorous inflammatory reaction when actinic keratoses are treated. It has the distinct advantage of identifying precancerous skin lesions not apparent on clinical inspection or palpation. Following a course of Efudex to the face, patients have been noted to have fewer signs of dermatoheliosis.

The investigators propose to determine if Efudex is associated with improvement of aging skin in the setting of treating actinic keratoses. The researchers hope to demonstrate less p53 staining following Efudex treatment. It is proposed that the skin improvements seen following a course of Efudex are due to both reduction of actinic keratoses and impact on photoaging. The researchers propose to quantify the effects of Efudex therapy on the immunohistochemical staining properties of facial skin with respect to p53 and procollagen. The hypothesis is that Efudex therapy will decrease p53 immunostaining thus providing biochemical evidence to support this treatment in the reduction of actinic keratoses with concomitant improvement of aging skin.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older of either gender.
* Patients must have actinic keratoses
* Patients must have clinical photoaging judged by rhytides, dyspigmentation, poikiloderma, lentigines, skin thinning, and/or telangiectases.
* Subjects must be in generally good health and willing to undergo skin biopsies from the face.
* Subjects must be willing and able to comply with the requirements of the protocol.
* You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* Oral retinoid therapy (such as Accutane) within two months of study entry.
* Topical retinoid, imiquimod, or diclofenac therapy within 2 months of study entry.
* Prior laser re-surfacing, chemical peels for actinic keratoses or aging skin.
* Pregnant or nursing subjects.
* Non-compliant subjects.
* Subjects with a significant medical history or concurrent illness that the investigator feels is not safe for study participation.
* Prior systemic treatment with 5-fluorouracil.
* Known history of allergy to lidocaine (numbing medication), 5-fluoruracil, or any other known components of Efudex.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Actinic Keratoses resolution and improvement in photoaging

SECONDARY OUTCOMES:
Changes in p53 immunostaining intensity will be used to assess response
Collagen production will be evaluated by Western blotting, immunohistology, and RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States